CLINICAL TRIAL: NCT03753789
Title: A Multicenter Study to Evaluate NEUWAVE Microwave Ablation System Using Ablation Confirmation in Patients With a Soft Tissue Liver Lesion
Brief Title: Ablation Confirmation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Combined study endpoints with ongoing registry (NOLA/NEU_2017_04)
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2017_03
Record Dates: First submitted 2018-10-31; First posted 2018-11-27 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cancer of the Liver; Liver Cancer; Neoplasms, Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microwave Ablation (Experimental): NEUWAVE Microwave Ablation System with AC software for patients undergoing a percutaneous ablation of a soft tissue liver lesion by an interventional radiologist.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Microwave Ablation — NEUWAVE microwave ablation of soft tissue liver lesions will be performed percutaneously by an interventional radiologist while the patient is under general anesthesia or deep conscious sedation.

SUMMARY:
Prospective, single-arm, multicenter study that will generate clinical data using the NEUWAVE MicroWave Ablation System with AC (Ablation Confirmation) software in patients undergoing ablation of a soft tissue liver lesion.

DETAILED DESCRIPTION:
Prospective, single-arm, multicenter study that will generate clinical data on 100 adult patients using the NEUWAVE MicroWave Ablation System with AC (Ablation Confirmation) software in patients undergoing ablation of a soft tissue liver lesion. AC software is a computed tomography (CT) image processing software package available as an optional feature for use with the NEUWAVE Microwave Ablation System. AC imports images from CT scanners for display and processing during ablation procedures to assist physicians in identifying ablation targets, assessing optimal ablation probe placement, and confirming the adequacy of the ablation margin.

All ablations will be performed percutaneously by an interventional radiologist while the patient is under general anesthesia or deep conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

1. A patient with at least one soft-tissue liver lesion less than or equal to 5cm undergoing microwave ablation using the NEUWAVE Microwave Ablation System. Note: a patient cannot have more than 3 lesions ablated during the procedure.
2. Intent to use Ablation Confirmation software (any AC software version permitted) during the ablation procedure.
3. Written Informed Consent to voluntarily participate in the study, follow CT scan schedule, and authorize the transfer of his/her data to the Sponsor
4. Patients greater than or equal to 22 years of age
5. Performance status 0-2 (Eastern Cooperative Oncology Group [ECOG]) classification
6. Class A or B functional hepatic reserve based on the Child-Pugh score.
7. Lesion must be visualized by non-contrast enhanced CT scan or the patient must tolerate contrast and meet institutional guidelines for contrast use based on glomerular filtration rate (GFR).

Exclusion Criteria:

1. Active bacterial infection or fungal infection on the day of the ablation.
2. Patients with implantable pacemakers or other electronic implants.
3. Platelet count less than 50,000/mm cubed.
4. Patients with uncorrectable coagulopathy at the time of ablation.
5. Currently breastfeeding or pregnant (latter confirmed by serum pregnancy test, per site's SOC).
6. Physical or psychological condition which would impair study participation.
7. ASA (American Society of Anesthesiologists) score of great or equal to 4.
8. Use of hydrodissection.
9. Systemic chemotherapy or radiation therapy for the liver, within 30 days prior to the study ablation procedure.
10. INR greater than 1.8.
11. Patient has participated in an investigational clinical study within 30 days of the screening visit for this study.
12. Patient judged unsuitable for study participation by the performing physician for any other reason.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Loma Linda University Medical Center, Loma Linda, California
  - UCLA, Los Angeles, California
  - Olives View - UCLA Medical Center, Sylmar, California
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 participants signed the informed consent, 7 of whom were later screen failures as they did not meet all inclusion/exclusion criteria. These 7 participants were not treated with the NEUWAVE microwave ablation device.
Pre-assignment Details: 39 participants met all inclusion/exclusion criteria. All participants were treated with the NEUWAVE microwave ablation device. However, 1 participant did not have the Ablation Confirmation software used in conjunction with the NEUWAVE microwave ablation device, as planned, and was therefore excluded in the full analysis set, defined as the 'Started' population.
Units Other Than Participants: Lesions
Groups:
- Microwave Ablation With Ablation Confirmation Software: Each participant underwent NEUWAVE microwave ablation using Ablation Confirmation software of at least one soft-tissue liver lesion in accordance with the study site's standard-of-care.
Period: Overall Study
Arm/Group | Microwave Ablation With Ablation Confirmation Software
Started (38) | 38; 47 Lesions (Signed the informed consent form, met all inclusion/exclusion criteria, and underwent NEUWAVE microwave ablation using the Ablation Confirmation software.)
Completed (36) | 36; 44 Lesions (Signed the informed consent form, met all inclusion/exclusion criteria, underwent NEUWAVE microwave ablation using the Ablation Confirmation software, and completed all follow-up study visits.)
Not Completed | 2; 3 Lesions
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Microwave Ablation With Ablation Confirmation Software
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (9.596)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 29
  Asian | 3
  Not Reported | 6
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 30.8 (5.469)
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 2
  Former Smoker | 15
  Non-Smoker | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lesions Where Probe Repositioning is Suggested
Time Frame: Day 0
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Microwave Ablation: Each participant underwent microwave ablation using NEUWAVE and the Ablation Confirmation software for at least one soft-tissue liver lesion in accordance with the study site's standard-of-care
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 38
Number analyzed (Lesions) | 47
Lesions
  Actions taken due to AC software indicating probe placement not satisfactory | 16
  No actions taken despite AC software indicating probe placement not satisfactory | 2
  No actions taken due to AC software indicating satisfactory probe placement | 29

2. Primary Outcome: Percentage of Lesions Where Re-ablation is Suggested
Time Frame: Day 0
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 38
Number analyzed (Lesions) | 47
Lesions
  Actions taken due to AC software indicating ablation margin not complete | 2
  No actions taken despite AC software indicating ablation margin not complete | 8
  No actions taken due to AC software indicating satisfactory margins | 37

3. Secondary Outcome: Technical Success
Description: Ablation of the target lesion(s) according to the protocol and covered completely with an adequate margin, as defined by the performing physician (that is, the ablation zone completely overlaps or encompasses the target lesion plus an adequate ablative margin)
Time Frame: Day 0
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 38
Number analyzed (Lesions) | 47
Lesions | 46

4. Secondary Outcome: Technique Efficacy
Description: Ablation of the target lesion(s) according to the protocol and covered completely with an adequate margin, as defined by the performing physician (that is, the ablation zone completely overlaps or encompasses the target lesion plus an adequate ablative margin) as assessed by imaging at 6 weeks
Time Frame: 6 weeks
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 38
Number analyzed (Lesions) | 44
Lesions | 44

5. Secondary Outcome: Hospital Resource Utilization
Description: How many days patients remain in the hospital after the ablation procedure
Time Frame: 6 weeks
Population: Only 27 patients had this data available. When not collected, this was noted as a protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 27
Participants
  Discharged the same day as the ablation procedure | 16
  Discharged after one night following the ablation procedure | 10
  Discharged two or more nights following the ablation procedure | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Per the study protocol, only events that the site investigator determined to be device-related and/or procedure-related were captured within the study database as this was a post-market study. These events were evaluated from the time of first probe puncture (Day 0) through study completion (6 weeks).
Arm/Group | Microwave Ablation With Ablation Confirmation Software
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation With Ablation Confirmation Software (N=38)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Perihepatic fluid collection (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation With Ablation Confirmation Software (N=38)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03753789/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03753789/SAP_001.pdf